CLINICAL TRIAL: NCT06814145
Title: A Phase 2, Multicenter, Double-blind, Extension Study to Evaluate the Effects of Sotatercept for the Treatment of Combined Postcapillary and Precapillary Pulmonary Hypertension (Cpc-PH) Due to Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Extension Study of Sotatercept in People With Pulmonary Hypertension (MK-7962-023)
Acronym: HARMONIZE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7962-023; MK-7962-023 (Other: MSD); U1111-1309-2142 (Registry Identifier: UTN); 2024-515773-99-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotatercept 0.3 mg/kg (Experimental): Participants receive sotatercept 0.3 mg/kg subcutaneous (SC) injection every 3 weeks (Q3W) for up to approximately 168 weeks or until discontinuation.
  Interventions: Biological: Sotatercept
- Sotatercept 0.7 mg/kg (Experimental): Participants receive sotatercept 0.7 mg/kg SC injection Q3W for up to approximately 168 weeks or until discontinuation.
  Interventions: Biological: Sotatercept

INTERVENTIONS:
Biological: Sotatercept — subcutaneous injection
  Other Names: ACE-011

SUMMARY:
Researchers are looking for new ways to treat people with a type of pulmonary hypertension called combined postcapillary and precapillary pulmonary hypertension (Cpc-PH). This study focuses on Cpc-PH that is caused by heart failure with preserved ejection fraction (HFpEF).

Researchers want to know if the study treatment, sotatercept, can treat people with Cpc-PH caused by HFpEF. This is an extension study, which means people who took part in a certain study on sotatercept for Cpc-PH (called a parent study) may be able to join this study. In this extension study, people will take sotatercept and researchers will follow their health for a longer time.

The main goal of this extension study is to learn about the long-term safety of sotatercept and if people tolerate it over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Completed MK-7962-007 (CADENCE) (Visit 9 and end of treatment [EOT] visit) without discontinuing study intervention and is able to safely enroll into MK-7962-007 (HARMONIZE)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a diagnosis of pulmonary hypertension (PH) in world health organization (WHO) Group 1, WHO Group 3, WHO Group 4, or WHO Group 5
* Has had a study intervention interruption
* Is pregnant or breastfeeding
* Has chronic liver disease with severe hepatic impairment and/or cirrhosis (eg, hepatic encephalopathy)
* Anticipation of more than 1 valve replacement or repair (mechanical or biomechanical) and/or have undergone more than 1 valve replacement or repair
* Has severe tricuspid regurgitation due to primary valvular disease (eg, from endocarditis, carcinoid, or mechanical destruction)
* Anticipated or undergone heart transplant or ventricular assist device implantation
* Has had prior exposure to luspatercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 187 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 168 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 48 | Baseline and Week 48
  PVR, a hemodynamic variable of pulmonary circulation, is measured by right heart catheterization (RHC). The change from baseline in PVR at Week 48 will be presented.
Change From Baseline in the 6-Minute Walk Distance (6MWD) at Week 48 | Baseline and Week 48
  The 6MWD tests the distance walked in 6 minutes as a measure of functional capacity. The change from baseline in 6MWD at Week 48 will be presented.
Change From Baseline in the 6MWD at Week 126 | Baseline and Week 126
  The 6MWD tests the distance walked in 6 minutes as a measure of functional capacity. The change from baseline in 6MWD at Week 126 will be presented.
Change From Baseline in the 6MWD at Week 174 | Baseline and Week 174
  The 6MWD tests the distance walked in 6 minutes as a measure of functional capacity. The change from baseline in 6MWD at Week 174 will be presented.
Change From Baseline in New York Heart Association Functional Class (NYHA FC) at Week 48 | Baseline and Week 48
  NYHA FC classifies the extent of heart failure. The change from baseline in NYHA FC at Week 48 will be presented.
Change From Baseline in NYHA FC at Week 126 | Baseline and Week 126
  NYHA FC classifies the extent of heart failure. The change from baseline in NYHA FC at Week 126 will be presented.
Change From Baseline in NYHA FC at Week 174 | Baseline and Week 174
  NYHA FC classifies the extent of heart failure. The change from baseline in NYHA FC at Week 174 will be presented.
Change From Baseline in N-terminal Pro-hormone Brain Natriuretic Peptide (NT-proBNP) at Week 48 | Baseline and Week 48
  NT-proBNP is an established marker of ventricular dysfunction in participants with PAH. NT-proBNP will be measured at baseline and at Week 48. The change from baseline in NT-proBNP at Week 48 will be presented.
Change From Baseline in NT-proBNP at Week 126 | Baseline and Week 126
  NT-proBNP is an established marker of ventricular dysfunction in participants with PAH. NT-proBNP will be measured at baseline and at Week 126. The change from baseline in NT-proBNP at Week 126 will be presented.
Change From Baseline in NT-proBNP at Week 174 | Baseline and Week 174
  NT-proBNP is an established marker of ventricular dysfunction in participants with PAH. NT-proBNP will be measured at baseline and at Week 174. The change from baseline in NT-proBNP at Week 174 will be presented.
Change From Week 24 in PVR at Week 48 | Week 24 and Week 48
  PVR, a hemodynamic variable of pulmonary circulation, is measured by right heart catheterization (RHC). The change from Week 24 in PVR at Week 48 will be presented.
Change From Week 24 in 6MWD at Week 48 | Week 24 and Week 48
  The 6MWD tests the distance walked in 6 minutes as a measure of functional capacity. The change from Week 24 in 6MWD at Week 48 will be presented.
Change From Week 24 in NYHA FC at Week 48 | Week 24 and Week 48
  NYHA FC classifies the extent of heart failure. The change from Week 24 in NYHA FC at Week 48 will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (54):
- United States (21):
  - Pulmonary Associates, PA ( Site 1008), Phoenix, Arizona
  - Jeffrey S. Sager, MD Medical Corporation ( Site 1060), Santa Barbara, California
  - Stanford University Medical Center ( Site 1024), Stanford, California
  - South Denver Cardiology Associates ( Site 1091), Littleton, Colorado
  - AdventHealth Orlando ( Site 1058), Orlando, Florida
  - The Emory Clinic ( Site 1030), Atlanta, Georgia
  - Norton Pulmonary Specialists ( Site 1066), Louisville, Kentucky
  - University Of Nebraska Medical Center ( Site 1053), Omaha, Nebraska
  - Weill Cornell Medical Center ( Site 1046), New York, New York
  - Duke University Medical Center ( Site 1026), Durham, North Carolina
  - The Carl and Edyth Lindner Center for Research and Education at the Christ Hospital ( Site 1001), Cincinnati, Ohio
  - The Cleveland Clinic Foundation. ( Site 1065), Cleveland, Ohio
  - The Ohio State University Wexner Medical Center ( Site 1032), Columbus, Ohio
  - Allegheny General Hospital ( Site 1088), Pittsburgh, Pennsylvania
  - Lankenau Medical Center ( Site 1089), Wynnewood, Pennsylvania
  - Rhode Island Hospital ( Site 1039), Providence, Rhode Island
  - Medical University of South Carolina ( Site 1003), Charleston, South Carolina
  - Statcare Pulmonary Consultants ( Site 1031), Knoxville, Tennessee
  - Intermountain Medical Center ( Site 1079), Murray, Utah
  - Inova Fairfax Medical Campus ( Site 1078), Falls Church, Virginia
  - Pulmonary Associates of Richmond - West Broad Street ( Site 1069), Richmond, Virginia
- Université Libre de Bruxelles - Hôpital Erasme ( Site 0100), Brussels, Bruxelles-Capitale, Region de, Belgium
- Hamilton Health Sciences Hamilton General Hospital ( Site 0004), Hamilton, Ontario, Canada
- France (6):
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur ( Site 0206), Nice, Alpes-Maritimes
  - Hopital Arnaud de Villeneuve ( Site 0200), Montpellier, Herault
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes ( Site 0205), Saint-Herblain, Loire-Atlantique
  - Centre Hopitalier Universitaire d'Angers ( Site 0204), Angers, Maine-et-Loire
  - CHU de Rouen ( Site 0203), Rouen, Seine-Maritime
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre ( Site 0202), Le Kremlin-Bicêtre, Val-de-Marne
- Germany (6):
  - Thoraxklinik-Heidelberg gGmbH ( Site 0309), Heidelberg, Baden-Wurttemberg
  - Krankenhaus Neuwittelsbach ( Site 0310), München, Bavaria
  - UKGM Gießen/Marburg ( Site 0312), Giessen, Hesse
  - Universitaetsklinikum Koeln ( Site 0311), Cologne, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz ( Site 0315), Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus Dresden ( Site 0301), Dresden, Saxony
- Israel (5):
  - Rambam Health Care Campus ( Site 0403), Haifa
  - Edith Wolfson Medical Center ( Site 0404), Holon
  - Hadassah Medical Center ( Site 0402), Jerusalem
  - Meir Medical Center ( Site 0401), Kfar Saba
  - ZIV Medical Center ( Site 0400), Safed
- Italy (3):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII ( Site 0502), Bergamo, Lombardy
  - Fondazione IRCCS Policlinico San Matteo ( Site 0501), Pavia
  - AOU Policlinico Umberto I ( Site 0500), Roma
- Unidad de Investigacion Clinica en Medicina, S.C. ( Site 2505), Monterrey, Nuevo León, Mexico
- Poland (3):
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II-Oddzial Kliniczny Chorob Serca i Naczyn z Podod ( Site 0600), Krakow, Lesser Poland Voivodeship
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego ( Site 0601), Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku ( Site 0603), Bialystok, Podlaskie Voivodeship
- Spain (5):
  - Hospital Costa del Sol ( Site 0704), Marbella, Malaga
  - Hospital Clinic I Provincial de Barcelona ( Site 0701), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 0702), Madrid
  - Hospital Universitario Virgen Macarena ( Site 0705), Seville
  - HOSPITAL GENERAL UNIVERSITARIO DE TOLEDO ( Site 0703), Toledo
- Sahlgrenska Universitetssjukhuset-Cardiology Research Unit ( Site 0800), Gothenburg, Västra Götaland County, Sweden
- Hammersmith Hospital-Department of Cardiology ( Site 0900), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com